CLINICAL TRIAL: NCT03516760
Title: A Multicenter, Open-label, Dose-escalating, Phase I Trial With GEM333, a CD33 Targeted Bispecific Antibody Engaging T-cells, in Relapsed or Refractory Acute Myeloid Leukemia
Brief Title: Dose-escalating Phase I Trial With GEM333 in Patients With Acute Myeloid Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The actions and measures to be taken to restart the trial could not be implemented which made the premature termination inevitability.
Sponsor: AvenCell Europe GmbH (Industry)
Collaborators: GCP-Service International Ltd. & Co. KG (Industry)
Responsible Party: Sponsor
Organization: AvenCell Therapeutics, Inc. (Industry)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GEM333-01; 2017-001707-77 (EudraCT Number)
Record Dates: First submitted 2018-04-06; First posted 2018-05-04 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Acute Myeloid Leukemia; Relapsed AML; Refractory AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Intervention Model Description: Dose escalation scheme; Single patient cohorts on the first three dose levels, 3+3 afterwards.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GEM333 (Experimental): application of GEM333, a CD33 targeted bispecific antibody engaging T-cells
  Interventions: Drug: GEM333

INTERVENTIONS:
Drug: GEM333 — infusion of GEM333; administered intravenously and continuously over 10 days

SUMMARY:
This dose-escalating phase I trial assesses for the first time the safety, the side effects and the harmlessness, as well as the therapeutical benefit of the new study drug GEM333 in patients with acute myeloid leukemia (AML). This AML was relapsed after previous therapy or was refractory to the standard therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients, ≥ 18 years of age
2. Documented definitive diagnosis of CD33 positive AML (according to standard of care testing) in

   * 2a. Patients having received standard induction chemotherapy: either refractory to standard induction treatment, or is relapsed within 6 months after achieving 1st CR, or relapsed later than 6 months after 1st CR and refractory to standard salvage regimen, or relapse after ≥ 2nd CR and not eligible for curative treatment (i.e. allogeneic stem cell transplantation)
   * 2b. Patients not eligible for standard induction chemotherapy: either refractory or progressive after at least 1 cycle of demethylating agents
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
4. Life expectancy of at least 2 months
5. Adequate renal and hepatic laboratory assessments:
6. Adequate cardiac function, i.e. left ventricular ejection fraction (LVEF) of ≥ 45% as assessed by transthoracal two-dimensional echocardiography
7. A female of childbearing potential may be enrolled providing she has a negative pregnancy test at screening visit and is routinely using a highly effective method of birth control (pearl index of ≤ 1 required) resulting in a low failure rate (e.g. hormonal contraception, intrauterine device, total sexual abstinence or sterilization) until 3 months from the last study drug administration. Male patients must also practice a highly effective method of birth control.
8. Able to give written informed consent
9. Weight ≥ 45 kg

Exclusion Criteria:

1. Acute promyelocytic leukemia (t15;17)
2. Manifestation of AML in central nervous system
3. Leukocytosis > 10 Gpt/L
4. Cardiac disease: i.e. heart failure NYHA III or IV; unstable coronary artery disease (Myocardial Infarction more than 6 months prior to study entry is permitted); serious cardiac ventricular arrhythmias requiring anti-arrhythmic therapy
5. Patients undergoing renal dialysis
6. Pulmonary disease with clinical relevant hypoxia (need for continuous oxygen inhalation)
7. Active central nervous diseases (e.g. parkinson, multiple sclerosis, epilepsy) and stroke within last 6 months
8. Active infectious disease considered by investigator to be incompatible with protocol
9. Allogeneic stem cell transplantation within last three months or GvHD requiring immune-suppressive therapy
10. Major surgery within 28 days prior to start of study medication
11. Other malignancy requiring active therapy but adjuvant endocrine therapy is allowed
12. Checkpoint inhibitors und CD33 targeting agents within 8 weeks prior to start of trial medication
13. Autoimmune diseases requiring systemic steroids or other systemic immunosuppressants
14. Treatment with any investigational drug substance or experimental therapy within 4 weeks prior to start of trial medication or 5 half lives of the substance prior to start of trial medication
15. Pregnant or breastfeeding women
16. Psychologic disorders, drug and/or significant active alcohol abuse
17. Known history of human immunodeficiency virus (HIV) or active/chronic infection with hepatitis C virus (HCV) or hepatitis B virus (HBV)
18. Known hypersensitivity to GEM333 excipients
19. Evidence suggesting that the patient is not likely to follow the study protocol (e.g. lacking compliance)
20. Incapability of understanding purpose and possible consequences of the trial
21. Patients who should not be included according to the opinion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-04-11 (Actual); Primary Completion 2022-06-14 (Actual); Study Completion 2022-06-14 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | End of Treatment (EOT) +8 days resp. +28 days (DLT period)
  MTD is the previous dose level of the cohort where a DLT is observed in at least wo subjects.
Incidence of dose limiting toxicity (DLT) | End of Treatment (EOT) +8 days resp. +28 days
  Dose Limiting Toxicity is defined as any event at least possibly related to IMP (complete definition provided protocol)
Incidence and intensity of adverse events graded according to CTCAE V4.03 | End of Treatment (EOT) +8 days resp. +28 days

SECONDARY OUTCOMES:
Recommended phase 2 dose | From start of treatment until up to +28 days after last treatment cycle (1 initial cycle + max. 2 additional cycles per patient). Each cycle consists of 10 days treatment plus DLT evaluation period (8 resp. 28 days, depending on blast clearance).
  The RP2D will be determined based on MTD, all available efficacy data, and all available safety data, including information derived from additional treatment cycles.
Complete remission (CR) | until two years after start of study medication
  bone marrow blasts < 5%, absence of extramedullary disease, absolute neutrophil count > 1 Gpt/L and platelet count > 100 Gpt/L
Composite complete remission (CRc) rate | until two years after start of study medication
  Rate at any time point, defined as the proportion of patients having either CR or CRi
Partial Remission (PR) | until two years after start of study medication
  All hematological criteria for CR with bone marrow blasts 5-25% and decrease of pre-treatment bone marrow blast percentage by at least 50 %.
Disease stabilization (DS) | until two years after start of study medication
  Reduction of blast percentage by 25% compared to baseline without normalization of peripheral blood counts to levels not qualifying for PR or CR
Best response rate | until two years after start of study medication
  Defined as the best observed response at any time point during observational period.
Duration of CRc | until two years after start of study medication
  Defined as the number of days between the date of CR/CRi achievement and the date of the last assessment confirming CR/CRi
Duration of PR | until two years after start of study medication
  Defined as the number of days between the date of PR achievement and the date of the last assessment confirming PR.
Progression free survival (PFS) | until two years after start of study medication
  Is defined as the time from first treatment with GEM333 until disease progression or death from any cause
Overall survival | until two years after start of study medication
  Defined as the number of days between the first study drug administration and death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Martin Wermke, MD, Principal Investigator — Universitätsklinikum Carl Gustav Carus Dresden
Locations (7):
- Germany (7):
  - Universitätsmedizin Mannheim, Mannheim, Baden-Wurttemberg
  - Klinikum rechts der Isar, München, Bavaria
  - Universitätsklinikum Würzburg, Würzburg, Bavaria
  - Universitätsklinikum Frankfurt, Frankfurt am Main, Hesse
  - Universitätsklinikum Marburg, Marburg, Hesse
  - Universitätsklinikum Dresden, Dresden, Saxony
  - Charité Universitätsmedizin, Berlin

IPD SHARING:
Plan to Share IPD: No